CLINICAL TRIAL: NCT01783483
Title: An Evaluation of Rigid Sternal Fixation in Supporting Bone Healing and Improving Postoperative Recovery: A Prospective, Randomized Trial
Brief Title: An Evaluation of Rigid Sternal Fixation in Supporting Bone Healing and Improving Postoperative Recovery
Acronym: SB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0712; SLBlu (Other: Biomet Microfixation)
Record Dates: First submitted 2013-01-31; First posted 2013-02-05 (Estimated); Results first posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-08

CONDITIONS: Coronary Artery Disease; Angina Pectoris; Cardiac Valve Disease
Keywords: CABG; Valve replacement; sternal closure; midline sternotomy; sternal plates
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Heart Valve Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suture Wire (Active Comparator): The closure technique should be per surgeon and institutional preference, with documentation of the wiring technique including the wiring configuration and number of wires used. A minimum of 6 wires that cross the midline sternotomy should be used (e.g. 6 simple wires, 3 double wires, 3 figure of 8 wires, etc.).
  Interventions: Device: Suture Wire
- SternaLock Blu closure system (Experimental): Patients will receive treatment option for sternal closure with the SternaLock Blue closure system at a minimum of 2 "X" plates on the sternal body and 1 "L" plate (or equivalent) on the manubrium. This technique is the standard configuration for this study, and is intended to ensure that at least 3 plates are used to achieve adequate fixation and stability, while allowing for variations in the plating configuration as a result of patient anatomy and surgeon preference. Various Sternal Blu plates may be used on the manubrium as described below, as can an additional plate on the sternal body.
  Interventions: Device: SternaLock Blue closure system

INTERVENTIONS:
Device: SternaLock Blue closure system — SternaLock Blue closure system is a primary closure system plate-based
  Other Names: SternaLock, SternalBlu
  Arms: SternaLock Blu closure system
Device: Suture Wire — Closure system wire-based used to approximate the two halfs of the sternum following a median sternotomy.
  Arms: Suture Wire

SUMMARY:
The primary objective of this study is to evaluate sternal bone healing following a full median sternotomy versus standard of care for sternal closure with wire cerclage. Additional outcomes on post-operative pain and analgesic usage, patient function and quality of life, and complications will also be collected. A health economics study will also be conducted, in which cost and billing data will be collected from sites participating in this clinical study.

DETAILED DESCRIPTION:
Rigid sternal fixation with the BIOMET SternaLock Blu Sternal Closure System may result in greater sternal stability that leads to superior sternal bone healing, less postoperative pain and narcotic usage, and improved functional outcomes compared to wire cerclage. The health economics analysis is an interesting component of this study, in which cost and billing data will be collected from participating sites and analyzed in terms of cost/effectiveness for patients and healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a full standard midline sternotomy as a result of a cardiac surgical procedure (i.e. coronary artery bypass graft (CABG) and/or valve replacement along with other cardiac surgical procedures)
* Patients admitted to the hospital the day of or the day before their scheduled surgical procedure
* Patients ≥ 18 years of age
* Patients with a BMI < 40

Exclusion Criteria:

Pre-operative

* Patients with endstage renal failure who are on dialysis
* Patients with severe chronic obstructive pulmonary disease (COPD) (FEV1 < 50% or patients on on-home oxygen)
* Patients on prescribed pre-operative narcotics
* Patients taking chronic steroids, biologics acting as immunosuppressants (e.g. Enbrel (etanercept), Humira (adalimumab), Remicade (infliximab), or chemotherapeutics (iv or oral chemotherapeutics for cancer). Patients using a steroid inhaler for asthma should not be excluded.
* Patients with an active infection as defined by a positive culture
* Patients with foreign body sensitivity
* Patients with mental or neurologic conditions who are unwilling or incapable of following postoperative care instructions
* Patients defined within the New York Heart Association (NYHA) or Canadian Cardiovascular Society (CCS) functional Class IV for congestive heart failure: i.e., patients with cardiac disease resulting in inability to carry on any physical activity without discomfort (CCS ; NYHA)
* Patients presenting emergent/salvage cardiac acuity as defined per the Society of Thoracic Surgeons (STS) guidelines: i.e., patients undergoing cardiopulmonary resuscitation en route to the operating room or prior to induction of anesthesia (STS)
* Patients unwilling or unable to return for follow-up

Operative

* Patients requiring delayed sternotomy closure
* Patients with an off-midline sternotomy reducing the bony margin between a SternaLock screw body and an osteotomy to within 2mm or less
* Patients presenting intra-operative conditions that in the opinion of the treating surgeon would require or preclude the use of either wire cerclage or rigid fixation, or who are not able to be plated or wired per the protocol (e.g. patients who in the opinion of the surgeon have insufficient quantity of quality of sternal bone; redo sternotomy with excessive fibrous tissue)
* Use of non resorbable (beeswax) bonewax
* Intraoperative death prior to device placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith B Allen, M.D., Principal Investigator — St Luke's Mid America and Vascular Institute
Locations (12):
- United States (12):
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Florida Hospital, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - United Heart & Vascular Clinic, United Hospital, part of Allina Health, Saint Paul, Minnesota
  - Saint Luke's Mid America Heart and Vascular Institute, Kansas City, Missouri
  - Columbia University Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - University of Toledo, Toledo, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Scott & White Memorial Hospital, Temple, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bennett-Guerrero E, Phillips-Bute B, Waweru PM, Gaca JG, Spann JC, Milano CA. Pilot study of sternal plating for primary closure of the sternum in cardiac surgical patients. Innovations (Phila). 2011 Nov;6(6):382-8. doi: 10.1097/IMI.0b013e318248fbda. PMID 22436774
- [Background] Casha AR, Yang L, Kay PH, Saleh M, Cooper GJ. A biomechanical study of median sternotomy closure techniques. Eur J Cardiothorac Surg. 1999 Mar;15(3):365-9. doi: 10.1016/s1010-7940(99)00014-7. PMID 10333037
- [Background] Chou SS, Sena MJ, Wong MS. Use of SternaLock plating system in acute treatment of unstable traumatic sternal fractures. Ann Thorac Surg. 2011 Feb;91(2):597-9. doi: 10.1016/j.athoracsur.2010.07.083. PMID 21256325
- [Background] Raman J, Lehmann S, Zehr K, De Guzman BJ, Aklog L, Garrett HE, MacMahon H, Hatcher BM, Wong MS. Sternal closure with rigid plate fixation versus wire closure: a randomized controlled multicenter trial. Ann Thorac Surg. 2012 Dec;94(6):1854-61. doi: 10.1016/j.athoracsur.2012.07.085. Epub 2012 Oct 25. PMID 23103010
- [Background] Hirose H, Yamane K, Youdelman BA, Bogar L, Diehl JT. Rigid sternal fixation improves postoperative recovery. Open Cardiovasc Med J. 2011;5:148-52. doi: 10.2174/1874192401105010148. Epub 2011 Jul 4. PMID 21760857
- [Background] Neaman KC, Blount AL, Kim JA, Renucci JD, Hooker RL. Prophylactic sternal plating with pectoralis advancement flaps after sternotomy in patients with a history of chest irradiation. Interact Cardiovasc Thorac Surg. 2011 Mar;12(3):355-8. doi: 10.1510/icvts.2010.247262. Epub 2010 Dec 7. PMID 21138917
- [Background] Snyder CW, Graham LA, Byers RE, Holman WL. Primary sternal plating to prevent sternal wound complications after cardiac surgery: early experience and patterns of failure. Interact Cardiovasc Thorac Surg. 2009 Nov;9(5):763-6. doi: 10.1510/icvts.2009.214023. Epub 2009 Aug 26. PMID 19710069
- [Background] Lee JC, Raman J, Song DH. Primary sternal closure with titanium plate fixation: plastic surgery effecting a paradigm shift. Plast Reconstr Surg. 2010 Jun;125(6):1720-1724. doi: 10.1097/PRS.0b013e3181d51292. PMID 20517097
- [Background] Shifrin DA, Sohn SM, Stouffer CW, Hooker RL, Renucci JD. Sternal salvage with rigid fixation in the setting of a massive mediastinal aortic pseudoaneurysm: a case report and review of the literature. J Plast Reconstr Aesthet Surg. 2008 Oct;61(10):e17-20. doi: 10.1016/j.bjps.2007.09.022. Epub 2007 Nov 26. PMID 18033747
- [Background] Raman J, Straus D, Song DH. Rigid plate fixation of the sternum. Ann Thorac Surg. 2007 Sep;84(3):1056-8. doi: 10.1016/j.athoracsur.2006.11.045. PMID 17720442
- [Background] Raman J, Song DH, Bolotin G, Jeevanandam V. Sternal closure with titanium plate fixation--a paradigm shift in preventing mediastinitis. Interact Cardiovasc Thorac Surg. 2006 Aug;5(4):336-9. doi: 10.1510/icvts.2005.121863. Epub 2006 Apr 25. PMID 17670585
- [Background] Dickie SR, Dorafshar AH, Song DH. Definitive closure of the infected median sternotomy wound: a treatment algorithm utilizing vacuum-assisted closure followed by rigid plate fixation. Ann Plast Surg. 2006 Jun;56(6):680-5. doi: 10.1097/01.sap.0000202825.41069.c3. PMID 16721085
- [Background] Song DH, Lohman RF, Renucci JD, Jeevanandam V, Raman J. Primary sternal plating in high-risk patients prevents mediastinitis. Eur J Cardiothorac Surg. 2004 Aug;26(2):367-72. doi: 10.1016/j.ejcts.2004.04.038. PMID 15296898
- [Background] Song DH, Agarwal JP, Jeevanandam V. Rigid sternal fixation in the cardiac transplant population. J Thorac Cardiovasc Surg. 2003 Sep;126(3):896-7. doi: 10.1016/s0022-5223(03)00605-6. No abstract available. PMID 14502187
- [Background] Pai S, Gunja NJ, Dupak EL, McMahon NL, Roth TP, Lalikos JF, Dunn RM, Francalancia N, Pins GD, Billiar KL. In vitro comparison of wire and plate fixation for midline sternotomies. Ann Thorac Surg. 2005 Sep;80(3):962-8. doi: 10.1016/j.athoracsur.2005.03.089. PMID 16122464
- See also: SternaLock Blu Primary Closure System Brochure — http://www.biomet.com/microfixation/getFile.cfm?id=3179&rt=inline
- See also: SternaLock Blu Product Description — http://www.biomet.com/microfixation/products.cfm?pdid=9&majcid=37&prodid=205

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were considered eligible for enrollment if they were undergoing an open heart surgery (e.g. CABG and/or valve surgery) with a full median sternotomy and met the inclusion/exclusion criteria. Patients were randomized at the time of sternal closure to receive either rigid sternal fixation (using sternal plates) or standard wire cerclage.
Period: Overall Study
Arm/Group | Suture Wire | SternaLock Blu Closure System
Started | 120 | 116
Completed | 100 | 101
Not Completed | 20 | 15
Not completed — Death | 3 | 3
Not completed — Lost to Follow-up | 14 | 10
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- SternaLock Blu Sternal Closure System: Patients will receive treatment option for sternal closure with the SternaLock Blue closure system at a minimum of 2 "X" plates on the sternal body and 1 "L" plate (or equivalent) on the manubrium. This technique is the standard configuration for this study, and is intended to ensure that at least 3 plates are used to achieve adequate fixation and stability, while allowing for variations in the plating configuration as a result of patient anatomy and surgeon preference. Various Sternal Blu plates may be used on the manubrium as described below, as can an additional plate on the sternal body.
  SternaLock Blue closure system: SternaLock Blue closure system is a primary closure system plate-based
- Total: Total of all reporting groups
Arm/Group | Suture Wire | SternaLock Blu Sternal Closure System | Total
Number analyzed (Participants) | 120 | 116 | 236
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.7 (11.4) | 65.3 (13.0) | 65.5 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 30 | 59
  Male | 91 | 86 | 177
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 102 | 103 | 205
  Black/African American | 12 | 7 | 19
  Hispanic/Latino | 5 | 4 | 9
  Asian | 0 | 1 | 1
  Not Given | 0 | 1 | 1
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 29.4 (4.6) | 28.8 (4.7) | 29.1 (4.7)
Risk Factor [Diabetes] [Count of Participants; unit: Participants] | 44 | 35 | 79
Risk Factor [Renal Failure] [Count of Participants; unit: Participants] | 2 | 0 | 2
Risk Factor [Current Cigarette Smoker] [Count of Participants; unit: Participants] | 10 | 14 | 24
Risk Factor [Hypertension] [Count of Participants; unit: Participants] | 83 | 86 | 169
Risk Factor [Chronic Lung Disease] [Count of Participants; unit: Participants]
  Mild | 15 | 18 | 33
  Moderate | 7 | 4 | 11
  Severe | 0 | 0 | 0
  None | 98 | 94 | 192
Risk Factor [Previous Sternotomy] [Count of Participants; unit: Participants] | 5 | 8 | 13
Risk Factor [Ejection Fraction] [Mean (Standard Deviation); unit: percentage] | 55.4 (11.3) | 55.2 (11.9) | 55.3 (11.6)
Risk Factor [Congestive Heart Failure by NYHA Classification] [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) classifies heart failure according to the severity of patients' symptoms. Grades I through 4 of heart failure by NYHA is a functional classification, placing patients in one of four categories based on how much they are limited during physical activity. Grade I represents better outcome since there is no limitation of physical activities while Grade IV (exclusionary for this trial) represents the worst outcome, since patients are unable to carry on any physical activity without discomfort, even at rest.
  Participants
    Class I - No limitation of physical activity | 17 | 10 | 27
    Class II - Slight limitation of physical activity | 27 | 21 | 48
    Class III - Marked limitation of physical activity | 11 | 15 | 26
    None (No heart failure present) | 65 | 70 | 135
Risk Factor [Peripheral Artery Disease] [Count of Participants; unit: Participants] | 5 | 12 | 17
Risk Factor [Cerebral Vascular Disease] [Count of Participants; unit: Participants] | 7 | 10 | 17
Risk Factor [Left Main Disease] [Count of Participants; unit: Participants] | 24 | 26 | 50
Risk Factor [Previous Myocardial Infarction] [Count of Participants; unit: Participants]
  More than 6h but less than 24h | 0 | 3 | 3
  More than 1 day but less than 7 days | 2 | 4 | 6
  More than 8 days but less than 21 days | 18 | 16 | 34
  More than 21 days | 0 | 1 | 1
  None or Never | 100 | 92 | 192
Inspirometry Volume [Mean (Standard Deviation); unit: mL] | 2436.3 (931.1) | 2398.7 (1025.7) | 2417.8 (976.8)

OUTCOME MEASURES:

1. Primary Outcome: Sternal Healing Score at 3 Month Post op, as Defined by a 6-point Scale to Evaluate Bone Healing
Description: Parameters for scoring:
  0 - Nonunion: No contact between sternal halves, absence of gap mineralization, and sclerotic osteotomy margins similar to that of cortical bone. Worst outcome
  1. - Indeterminate: No contact or mineralization between the sternal halves, but osteotomy margins were nonsclerotic, concave, or irregular
  2. - Early healing: Faint mineralization between noncontacting sternal halves, or a thin (1 mm) bridge of bone connecting the sternal halves anteriorly or posteriorly, or near bone-on-bone contact between the sternal halves, with sclerotic osteotomy margins
  3. - Mild synthesis: Bridging bone (i.e., no perceptible gap) along less than 50% of the anteroposterior dimension of the sternal halves, with the sternal halves either offset in the anteroposterior dimension, or aligned in the anteroposterior dimension
  4. - Moderate synthesis: Bridging bone along 50% or more of the antero-posterior dimension of the sternal haves 5- Sternal halves well-aligned. Best outcome
Time Frame: 3-month post-op
Population: Subjects with completed CT scan at 3 month post op: 102 Suture Wire / 103 SternaLock Blu
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Suture Wire | SternaLock Blu Closure System
Number analyzed (Participants) | 102 | 103
units on a scale | 1.8 (1.0) | 2.6 (1.1)
Statistical Analysis 1: Comparison: Suture Wire vs SternaLock Blu Closure System; Comparison of mean CT scan scores; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

2. Primary Outcome: Sternal Healing Score at 6 Month Post op, as Defined by a 6-point Scale to Evaluate Bone Healing
Description: Parameters for scoring:
  0 - Nonunion: No contact between sternal halves, absence of gap mineralization, and sclerotic osteotomy margins similar to that of cortical bone. Worst outcome
  1. - Indeterminate: No contact or mineralization between the sternal halves, but osteotomy margins were non-sclerotic, concave, or irregular
  2. - Early healing: Faint mineralization between non-contacting sternal halves, or a thin (1 mm) bridge of bone connecting the sternal halves anteriorly or posteriorly, or near bone-on-bone contact between the sternal halves, with sclerotic osteotomy margins
  3. - Mild synthesis: Bridging bone (i.e., no perceptible gap) along less than 50% of the anteroposterior dimension of the sternal halves, with the sternal halves either offset in the anteroposterior dimension, or aligned in the anteroposterior dimension
  4. - Moderate synthesis: Bridging bone along 50% or more of the anteroposterior dimension of the sternal haves 5- Sternal halves well-aligned. Best outcome
Time Frame: 6-month post-op
Population: Subjects with completed CT scan at 6 months post op: 100 Suture Wire / 101 SternaLock Blu)
Measure: Mean (Standard Deviation); unit: units on a scale 0-5
Arm/Group | Suture Wire | SternaLock Blu Closure System
Number analyzed (Participants) | 100 | 101
units on a scale 0-5 | 3.3 (1.1) | 3.8 (1.0)
Statistical Analysis 1: Comparison: Suture Wire vs SternaLock Blu Closure System; Test type: Superiority or Other; p = 0.0007, t-test, 2 sided

3. Secondary Outcome: Pain Measured in a 10-point Scale at Day 7 Post Operative
Description: Intensity of sternal pain assessed using 10 point scale:
  1. At rest
  2. After forced coughing. Patients score pain 0 to 10 where 0 represents no pain and 10 represents the worst pain a patient can experience
Time Frame: Day 7
Population: Pain assessed at resting and after forced coughing. Pain levels of 1 or more were deemed to have pain.
  Subjects at 7-Day post op with completed pain assessment: 31 Suture Wire / 30 SternaLock Blu
Measure: Mean (Standard Deviation); unit: units on a scale 0-10
Arm/Group | Suture Wire | SternaLock Blu Closure System
Number analyzed (Participants) | 31 | 30
units on a scale 0-10
  At Rest | 2.10 (2.52) | 1.07 (1.41)
  After Forced Coughing | 4.23 (2.64) | 2.20 (2.06)
Statistical Analysis 1: Comparison: Suture Wire vs SternaLock Blu Closure System; At Rest; Test type: Superiority or Other; p = 0.0539, t-test, 2 sided
Statistical Analysis 2: Comparison: Suture Wire vs SternaLock Blu Closure System; After Forced Coughing; Test type: Superiority or Other; p = 0.0015, t-test, 2 sided

4. Secondary Outcome: Pain Measured in a 10-point Scale at 3-week Post Operative
Description: Intensity of sternal pain assessed using 10 point scale in the following circumstances:
  1. At rest
  2. After forced coughing. Patients score pain 0 to 10 where 0 represents no pain and 10 represents the worst pain a patient can experience
Time Frame: 3-week Post-op
Population: Pain assessed at resting and after forced coughing. Only patients who reported pain levels of 1 or more were deemed to have pain.
  Subjects at 3-week post op with completed pain assessment: 107 Suture Wire / 107 SternaLock Blu
Measure: Mean (Standard Deviation); unit: units on a scale 0-10
Arm/Group | Suture Wire | SternaLock Blu Closure System
Number analyzed (Participants) | 107 | 107
units on a scale 0-10
  At Rest | 1.04 (1.57) | 0.79 (1.37)
  After Forced Coughing | 2.99 (2.56) | 1.92 (2.30)
Statistical Analysis 1: Comparison: Suture Wire vs SternaLock Blu Closure System; At Rest; Test type: Superiority or Other; p = 0.2125, t-test, 2 sided
Statistical Analysis 2: Comparison: Suture Wire vs SternaLock Blu Closure System; After Forced Coughing; Test type: Superiority or Other; p = 0.0014, t-test, 2 sided

5. Secondary Outcome: Pain Measured in a 10-point Scale at 6-week Post Operative
Description: as for outcome 4
Time Frame: 6-week Post-op
Population: Pain assessed at resting and after forced coughing. Only patients who reported pain levels of 1 or more were deemed to have pain.
  Subjects at 6-week post op with completed pain assessment: 114 Suture Wire / 112 SternaLock Blu
Measure: Mean (Standard Deviation); unit: units on a scale 0-10
Arm/Group | Suture Wire | SternaLock Blu Closure System
Number analyzed (Participants) | 114 | 112
units on a scale 0-10
  At Rest | 1.14 (1.91) | 0.54 (1.15)
  After Forced Coughing | 1.90 (2.19) | 1.26 (1.88)
Statistical Analysis 1: Comparison: Suture Wire vs SternaLock Blu Closure System; At Rest; Test type: Superiority or Other; p = 0.0049, t-test, 2 sided
Statistical Analysis 2: Comparison: Suture Wire vs SternaLock Blu Closure System; After Forced Coughing; Test type: Superiority or Other; p = 0.0183, t-test, 2 sided

6. Secondary Outcome: Pain Measured in a 10-point Scale at 3-month Post Operative
Description: as for outcome 4
Time Frame: 3-month Post-op
Population: Pain assessed at resting and after forced coughing. Pain levels of 1 or more were deemed to have pain.
  Subjects at 3-month post op with completed pain assessment 108 Suture Wire / 105 SternaLock Blu
Measure: Mean (Standard Deviation); unit: units on a scale 0-10
Arm/Group | Suture Wire | SternaLock Blu Closure System
Number analyzed (Participants) | 108 | 105
units on a scale 0-10
  At Rest | 0.46 (1.03) | 0.39 (1.38)
  After Forced Coughing | 1.01 (1.73) | 0.74 (1.49)
Statistical Analysis 1: Comparison: Suture Wire vs SternaLock Blu Closure System; At Rest; Test type: Superiority or Other; p = 0.6653, t-test, 2 sided
Statistical Analysis 2: Comparison: Suture Wire vs SternaLock Blu Closure System; After Forced Coughing; Test type: Superiority or Other; p = 0.2295, t-test, 2 sided

7. Secondary Outcome: Pain Measured in a 10-point Scale at 6-month Post Operative
Description: as for outcome 4
Time Frame: 6-month Post-op
Population: Pain assessed at resting and after forced coughing. Pain levels of 1 or more were deemed to have pain.
  Subjects at 6-month post op with completed pain assessment: 96 Suture Wire / 102 SternaLock Blu
Measure: Mean (Standard Deviation); unit: units on a scale 0-10
Arm/Group | Suture Wire | SternaLock Blu Closure System
Number analyzed (Participants) | 96 | 102
units on a scale 0-10
  At Rest | 0.65 (1.38) | 0.55 (1.43)
  After Forced Coughing | 0.76 (1.56) | 0.54 (1.26)

8. Secondary Outcome: Narcotic Usage
Description: Narcotics usage was tabulated and recorded at each follow-up interval and converted to Morphine Equivalence Dose (MED).
Time Frame: Index (Day 0 to Hospital Discharge)
Population: Subjects with completed narcotic usage assessment from Day 0 to hospital discharge: 118 Suture Wire / 114 SternaLock Blu
Measure: Mean (Standard Deviation); unit: milligrams of Morphine Equivalence Dose
Arm/Group | Suture Wire | SternaLock Blu Closure System
Number analyzed (Participants) | 118 | 114
milligrams of Morphine Equivalence Dose | 72.75 (104.02) | 93.73 (227.28)
Statistical Analysis 1: Comparison: Suture Wire vs SternaLock Blu Closure System; Index (Day 0 to Hospital Discharge); Test type: Superiority or Other; p = 0.370, t-test, 2 sided

9. Secondary Outcome: Narcotic Usage
Description: Narcotics usage was tabulated and recorded at each follow-up interval and converted to Morphine Equivalence Dose (MED) .
Time Frame: From Hospital Discharge to 3-week post-op
Population: Subjects with completed narcotic usage assessment from hospital discharge to 3-week post op: 109 Suture Wire / 112 SternaLock Blu
Measure: Mean (Standard Deviation); unit: milligrams of Morphine Equivalence Dose
Arm/Group | Suture Wire | SternaLock Blu Closure System
Number analyzed (Participants) | 109 | 112
milligrams of Morphine Equivalence Dose | 33.04 (61.82) | 29.65 (110.28)
Statistical Analysis 1: Comparison: Suture Wire vs SternaLock Blu Closure System; From Hospital Discharge to 3-week; Test type: Superiority or Other; p = 0.778, t-test, 2 sided

10. Secondary Outcome: Narcotic Usage
Description: Narcotics usage was tabulated and recorded at each follow-up interval and converted to Morphine Equivalence Dose (MED) .
Time Frame: From 3-week to 6-week post-op
Population: Subjects with completed narcotic usage assessment from 3-week to 6-week post op: 115 Suture Wire / 111 SternaLock Blu
Measure: Mean (Standard Deviation); unit: milligrams of Morphine Equivalence Dose
Arm/Group | Suture Wire | SternaLock Blu Closure System
Number analyzed (Participants) | 115 | 111
milligrams of Morphine Equivalence Dose | 9.65 (35.18) | 3.04 (9.92)
Statistical Analysis 1: Comparison: Suture Wire vs SternaLock Blu Closure System; From 3-week to 6-week post-op; Test type: Superiority or Other; p = 0.055, t-test, 2 sided

11. Secondary Outcome: Narcotic Usage
Description: Narcotics usage was tabulated and recorded at each follow-up interval and converted to Morphine Equivalence Dose (MED) .
Time Frame: From 6-week to 3-month post-op
Population: Subjects with completed narcotic usage assessment from 6-week to 3-month post op: 108 Suture Wire / 104 SternaLock Blu
Measure: Mean (Standard Deviation); unit: milligrams of Morphine Equivalence Dose
Arm/Group | Suture Wire | SternaLock Blu Closure System
Number analyzed (Participants) | 108 | 104
milligrams of Morphine Equivalence Dose | 17.11 (120.80) | 5.32 (25.08)

12. Secondary Outcome: Narcotic Usage
Description: Narcotics usage was tabulated and recorded at each follow-up interval and converted to Morphine Equivalence Dose (MED) .
Time Frame: From 3-month to 6 month post-op
Population: Subjects with completed narcotic usage assessment from 3-month to 6-month post op: 100 Suture Wire / 102 SternaLock Blu
Measure: Mean (Standard Deviation); unit: milligrams of Morphine Equivalence Dose
Arm/Group | Suture Wire | SternaLock Blu Closure System
Number analyzed (Participants) | 100 | 102
milligrams of Morphine Equivalence Dose | 48.32 (282.77) | 3.00 (12.72)
Statistical Analysis 1: Comparison: Suture Wire vs SternaLock Blu Closure System; From 3 month to 6-month post op; Test type: Superiority or Other; p = 0.113, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From Day 0 to 6-month post op.
Description: Serious Adverse Events reporting sternal wound complications, deaths, bleeding requiring re-operations, stroke and acute renal failure per patient from Day 0 to 6-month post op. Other Adverse Events are reported if frequency of occurrence was higher than 5%
Arm/Group | Suture Wire | SternaLock Blu Closure System
All-Cause Mortality (participants affected / at risk) | 3/120 | 2/116
Serious Adverse Events (participants affected / at risk) | 10/120 | 2/116
Other Adverse Events (participants affected / at risk) | 40/120 | 37/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suture Wire (N=120) | SternaLock Blu Closure System (N=116)
Deep Sternal Wound Infection (DSWI) (Infections and infestations) | 3 (8) | 0 (0) — DSWI must meet all of the following: * Wound opened with excision of tissue (I&D) or re-exploration of mediastinum * Positive culture unless patient on antibiotics or no culture obtained * Treatment with antibiotics beyond perioperative prophylaxis
Superficial Sternal Wound Infection (SSWI) (Infections and infestations) | 2 (2) | 0 (0) — Sternal Wound Infections not meeting criteria for DSWI
Other Sternal Wound Complication (Surgical and medical procedures) | 1 (1) | 0 (0) — Sternal complications not related to infection (i.e., pain requiring hardware removal)
Bleeding requiring re-operation (Cardiac disorders) | 2 (2) | 2 (2)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Acute Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suture Wire (N=120) | SternaLock Blu Closure System (N=116)
Arrythmia (Cardiac disorders) | 40 (40) | 37 (37)

LIMITATIONS AND CAVEATS:
At closing of this study, only 2 prospective RCTs have been conducted that compare RPF with WC. Because both were done with first and second generation devices from the same manufacturer, conclusions on the class effect of RPF systems cannot be made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No